CLINICAL TRIAL: NCT04193735
Title: A Case-control Study of the Gastrointestinal Response to a Liquid Test Meal in Chronic Intestinal Pseudo-obstruction, Using Magnetic Resonance Imaging
Brief Title: Pseudo-obstruction Assessment With MRI
Acronym: POM
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Pseudo-Obstruction Research Trust (Unknown); Northern Care Alliance NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); Cambridge University Hospitals NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Barts & The London NHS Trust (Other); London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19069
Record Dates: First submitted 2019-11-22; First posted 2019-12-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Chronic Intestinal Pseudo-Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIPO (case): MRI scan of gastrointestinal content and activity
  Interventions: Diagnostic Test: MRI scans after a liquid meal
- Chronic constipation (control): MRI scan of gastrointestinal content and activity
  Interventions: Diagnostic Test: MRI scans after a liquid meal

INTERVENTIONS:
Diagnostic Test: MRI scans after a liquid meal — Participants will be scanned fasted, then receive a liquid meal, then be scanned every half hour, seven times

SUMMARY:
This study will explore the potential for a standardized MRI scan after a liquid meal to be used in diagnosis of the rare but debilitating chronic intestinal pseudo-obstruction (CIPO).

DETAILED DESCRIPTION:
People with chronic intestinal pseudo-obstruction (CIPO) have problems digesting their food properly, due to a problem in their gut nerves or muscle. There are not many good tests to assess how a patient's stomach and bowels are working. Finding out more is the first step in developing a standardized clinical test using MRI to provide a faster diagnosis than is currently possible. Magnetic resonance imaging (MRI) scans allow the investigators to see inside the abdomen. Scans are not painful or harmful and are therefore ideal for repeated measurements. By scanning participants both before and after a test drink the investigators can see exactly how their digestion is working.

The investigators are inviting 16 people who are at least 16 years old, 8 who have CIPO and 8 with chronic constipation, so the investigators can compare the images. Participants will come in for one half day of scanning. The investigators will take a total of 8 scans of their abdomens, every half hour. Participants will also fill in symptom questionnaires at every scan, for example if they feel bloated or have any abdominal pain. Each scan will take about 15 minutes and will require short breath holds. Participants will be able to get out of the scanner at any time point if they feel the need to.

Participants will arrive fasted in the morning and will receive a test drink (a milk-based drink used as an oral nutritional supplement) right after the first scan. All participants will be asked to pause some of their usual medication that has a direct influence on digestion for 24h before the scan day and during the ~4h of the study.

The primary outcome is peak small bowel motility, which the investigators hypothesize to be less active in people with CIPO. Other outcomes include gastric volume, small bowel water content and distribution, peak gastric motility, and gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Sufficient level of English language to understand study information and respond to symptom questionnaires
* CASES: a clinical diagnosis of primary or secondary Chronic Intestinal Pseudo-Obstruction, excluding adhesional obstruction. PICs will be asked to send clinical documentation that the diagnosis has been confirmed on crosssectional imaging.
* CONTROLS: a Chronic constipation disorder diagnosed according to Rome IV criteria for functional constipation, constipation-predominant irritable bowel syndrome or opioid-induced constipation (diagnostic criteria as listed in Lacy et al 2016)

Exclusion Criteria:

* Inability to tolerate 400 ml liquid challenge meal (oral or through established gastrostomy; according to self-assessment)
* Contra-indication to MRI scanning, such as metal implants, pacemaker etc
* Pregnancy declared by candidate (no formal testing)
* Inability to stop short-acting medications likely to alter small bowel motility, such as antiemetics, fast release opioids, laxatives, and anti-diarrhoeals, on the day before the study (24h before baseline scan; i.e. a total of circa 30h) as well as antibiotics for three days before the study. This only applies to long-term antibiotics commonly given for dysbiosis (small intestinal bacterial overgrowth). A short course of antibiotics given for acute infections will not be interrupted but the study day will be delayed until the course is finished. Patches, long acting formulations such as slow release medication or depot injection medication will be allowed to continue
* Inability to omit parenteral nutrition for 12 hours before the fasting MRI scan (~16h total)
* Medical comorbidity that means subject will not be able to undergo multiple scans e.g. severe respiratory disorder limiting time lying flat; severe musculoskeletal disorder limiting mobility
* Previous small bowel resection (excluding ileostomy, insertion of venting tube or percutaneous endoscopic gastrostomy, appendectomy or cholecystectomy). Patients who have had a colectomy for their CIPO will be eligible.
* Other gastrointestinal disorder likely to alter small bowel function e.g. uncontrolled coeliac disease, Crohn's disease. A diagnosis of small intestinal bacterial overgrowth will not be a reason for exclusion. PICs will be asked to supply information on resections and comorbidities for CIPO participants.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases will be recruited through Digestive Diseases clinical services across England; Controls will be recruited from the population of Nottingham.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak small gut motility after a test liquid meal | up to 3.5 hours after meal, measured every half hour
  Investigating whether people with CIPO have a lower peak small gut motility after a test drink than people who do not have CIPO. Small gut motility will be assessed with a standardised method on CineMRI, based on power spectrum analysis of voxel-signal changes with time (the outcome will be reported in arbitrary units). The primary outcome is peak small gut motility since a delay in motility (linked to one specific time point) would not be sufficient to explain the difference between CIPO and controls.

SECONDARY OUTCOMES:
Gastric emptying rate (ml/min) after a test liquid meal | up to 3.5 hours after meal, measured every half hour
  Investigating whether people with CIPO have slower gastric emptying after a test drink than people who do not have CIPO. The gastric emptying rate is determined by measuring the gastric volume every half hour after the standardised meal.
Small bowel water volume (ml) after a test liquid meal | up to 3.5 hours after meal, measured every half hour
  Investigating whether people with CIPO have a greater volume of small bowel water after a test drink than people who do not have CIPO. Small bowel water content is determined from a heavily T2-weighted scan. The intensity threshold for free water will be set using each participant's spinal fluid, and only small bowel contents having an intensity equal to or greater than this value will be measured as small bowel free water volume.
Gastric motility after a test liquid meal | up to 3.5 hours after meal, measured every half hour
  Investigating whether people with CIPO have a reduced gastric motility after a test drink than people who do not have CIPO. Gastric motility will be assessed with a standardised method on CineMRI, based on power spectrum analysis of voxel-signal changes with time (the outcome will be reported in arbitrary units).

CONTACTS AND LOCATIONS:
Overall Officials: Giles Major, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised IPD may be available for sharing as part of collaborative data pooling but will not automatically be published as open source due to the possibility of identification through meta-data in a rare disease.